CLINICAL TRIAL: NCT06695845
Title: A Phase 2, Open-label, Multicenter Study to Evaluate Efficacy and Safety of Zanidatamab for the Treatment of Participants With Previously Treated HER2-expressing Solid Tumors (DiscovHER PAN-206)
Brief Title: A Phase 2 Study of Zanidatamab in Patients With HER2-expressing Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Jazz Pharmaceuticals Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JZP598-206; 2024-516551-41-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Gastric Cancer; Esophageal Cancer; Gastroesophageal Cancer; Colorectal Cancer; Endometrial Cancer; Non-small Cell Lung Cancer; Ovarian Cancer; Urothelial Carcinoma; Salivary Gland Cancer; Pancreatic Cancer; HER-2 Protein Overexpression
Keywords: JZP598; ZW25; HER2 IHC 3+ Overexpression Solid Tumors
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Carcinoma, Transitional Cell; Salivary Gland Neoplasms; Pancreatic Neoplasms | interventions — zanidatamab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanidatamab treatment arm (Experimental): Eligible participants receiving zanidatamab treatment
  Interventions: Drug: Zanidatamab

INTERVENTIONS:
Drug: Zanidatamab — Administered by intravenous (IV) infusion
  Other Names: ZW25; JZP598; ZIIHERA®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of zanidatamab for the treatment of participants with previously treated solid tumors that have Human Epidermal Growth Factor Receptor 2 (HER2) Immunohistochemistry (IHC) 3+ overexpression.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age inclusive at the time of signing the informed consent
2. Participants with locally advanced, unresectable, or metastatic solid tumors (except Biliary Tract Cancer (BTC), defined as gallbladder cancer or cholangiocarcinoma) who have progressed following at least 1 prior systemic treatment for metastatic or advanced disease and have no available treatment options that have confirmed benefit. Prior treatment with HER2-targeted therapy is not permitted (Cohort 1 only). For participants with breast cancer (Cohort 2) or GEA (Cohort 3), prior HER2-targeted therapy is permitted and prior therapy with trastuzumab deruxtecan (T-DXd) is required.
3. HER2 overexpression (IHC 3+) must be determined by a sponsor designated central laboratory.
4. All participants must have adequate tumor sample for submission to allow central HER2 testing.
5. Presence of at least 1 measurable lesion as assessed by Independent Central Review (ICR) based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
6. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Has a life expectancy of at least 3 months, in the opinion of the investigator.
8. Participants with history of treated and stable CNS metastases are eligible, provided the following criteria are met:

   1. Participants also have measurable metastatic disease with HER2 overexpression (IHC 3+) outside the CNS.
   2. Participants with treated CNS metastases that are no longer symptomatic may be included in the study if they recovered to < Grade 1 (CTCAE Version 5.0 or higher) or baseline from the acute toxic effect associated with the treatment > 7 days prior to Cycle 1 Day 1.
   3. Prior stereotactic radiosurgery or stereotactic radiotherapy should be completed at least 7 days (≥ 7 days) before the first dose of study intervention.
9. Adequate organ functions.
10. Females of childbearing potential must have a negative pregnancy test result.
11. Females of childbearing potential and males with a partner of childbearing potential must be willing to use 2 methods of birth control.

Exclusion Criteria:

1. Has known or suspected leptomeningeal disease and/or untreated brain metastasis.
2. Has uncontrolled or significant cardiovascular disease
3. Has ongoing toxicity related to prior cancer therapy
4. Has uncontrolled infection or requiring IV antibiotics, antivirals, or antifungals.
5. Has known Human Immunodeficiency Virus (HIV) infection.
6. Has active hepatitis B or C infection.
7. Has an active SARS-CoV-2 infection.
8. Has a history of life-threatening hypersensitivity to monoclonal antibody (mAbs) or to recombinant proteins or excipients in the drug formulation of zanidatamab.
9. Has any serious underlying medical or psychiatric condition that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site.
10. Has any issue or condition that, in the opinion of the investigator, would contraindicate the participant's participation in the study or confound the results of the study.
11. Prior treatment with HER2-targeted therapy (Cohort 1 only).
12. Has a history of trauma or major surgery
13. Was treated with systemic antineoplastic therapy, including hormonal therapies for breast cancer, or any investigational therapy within 4 weeks or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
14. Received zanidatamab at any time prior to the current study.
15. Colorectal Cancer (CRC) participants with known KRAS/NRAS and BRAF mutations.
16. Non-Small Cell Lung Cancer (NSCLC) participants with known ALK, EGFR mutations and ROS1 fusion.
17. Female participants who are breastfeeding or pregnant, and female and male participants planning a pregnancy.
18. Prior or concurrent invasive malignancy other than the disease under study, whose natural history or treatment has, in the opinion of the investigator or medical monitor, the potential to interfere with the safety or efficacy assessment of the investigational regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (cORR) per RECIST Version 1.1, as assessed by ICR | Up to 2.5 years
  The Independent Central Review (ICR) assessed cORR is defined as the proportion of participants who had a best overall response of Complete Response (CR), or Partial Response (PR) based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Duration of Response (DOR) Per RECIST Version 1.1, as assessed by ICR | Up to 2.5 years
  ICR assessed DOR is defined as the time in months from the first objective response (CR or PR) that is subsequently confirmed to documented progressive disease (PD) per RECIST v1.1 or death from any cause.
cORR by RECIST Version 1.1, as assessed by Investigator | Up to 2.5 years
  Investigator assessed cORR is defined as the proportion of participants who had a best overall response of Complete Response (CR), or Partial Response (PR) based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Duration of Response (DOR) Per RECIST Version 1.1, as assessed by Investigator | Up to 2.5 years
  Investigator assessed DOR is defined as the time in months from the first objective response (CR or PR) that is subsequently confirmed to documented progressive disease (PD) per RECIST v1.1 or death from any cause.
Time to Response (TTR), as assessed by ICR | Up to 2.5 years
  ICR assessed TTR is defined as the time from the first dosing date to the first objective response (CR or PR) per RECIST v1.1.
Time to Response (TTR), as assessed by Investigator | Up to 2.5 years
  Investigator assessed TTR is defined as the time from the first dosing date to the first objective response (CR or PR) per RECIST v1.1.
Disease control rate (DCR), as assessed by ICR | Up to 2.5 years
  ICR assessed DCR is defined as the proportion of participants whose best overall response (BOR) is confirmed CR, or PR, or stable disease using the RECIST version 1.1 criteria
Disease control rate (DCR), as assessed by Investigator | Up to 2.5 years
  Investigator assessed DCR is defined as the proportion of participants whose best overall response (BOR) is confirmed CR, or PR, or stable disease using the RECIST version 1.1 criteria
Progression Free Survival (PFS), as assessed by ICR | Up to 2.5 years
  PFS is defined as the time in months from the first dosing date to the date of first documented disease progression (as assessed by ICR according to RECIST v1.1) or death from any cause, whichever occurs first.
Progression Free Survival (PFS), as assessed by Investigator | Up to 2.5 years
  PFS is defined as the time in months from the first dosing date to the date of first documented disease progression (as assessed by Investigator according to RECIST v1.1) or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 3.5 years
  OS is defined as the time in months from randomization to the date of death due to any cause.
Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) As Graded by NCI CTCAE Version 5.0 | Up to 2.5 years
Number of Participants With Dose Reductions | Up to 2.5 years
Number of Participants Discontinuing Study Treatment Due to TEAEs | Up to 2.5 years
Serum Concentrations of Zanidatamab | Up to 2.5 years
Number of Participants Positive for Anti-drug Antibodies to Zanidatamab | Up to 2.5 years
Number of participants reporting Symptomatic Adverse Events based on Patient-reported Outcome-Common Terminology Criteria for AEs (PRO-CTCAE) | Up to 2.5 years
Number of participants reporting Symptomatic Adverse Events based on European Organisation for Research and Treatment of Cancer (EORTC) Item Library | Up to 2.5 years
Percentage of all treated participants reporting overall side-effect bother on the Functional Assessment of Chronic Illness Therapy General Physical Item 5 (FACIT-GP5) | Up to 2.5 years
Percentage of time when participants on treatment reported a high side-effect bother on the Functional Assessment of Chronic Illness Therapy General Physical Item 5 (FACIT-GP5) | Up to 2.5 years

CONTACTS AND LOCATIONS:
Locations (21):
- United States (16):
  - Arizona Oncology Associates, PC - NAHOA, Prescott, Arizona
  - Rocky Mountain Cancer Center, Littleton, Colorado
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - Lake Nona, Orlando, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - Affiliated Oncologists, Chicago Ridge, Illinois
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Alliance Cancer Specialists, Horsham, Pennsylvania
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - West Texas, Amarillo, Texas
  - Texas Oncology - DFW, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Blue Ridge Cancer Care, Roanoke, Virginia
- South Korea (5):
  - Samsung Medical Center, Gangnam-gu, Seoul
  - Seoul National University Hospital, Jongno-gu, Seoul
  - Severance Hospital, Seodaemun-gu, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com.
URL: https://www.jazzpharma.com/science/clinical-trial-data-sharing